CLINICAL TRIAL: NCT02896088
Title: Prevention of Dental Caries in Primary Molars on Sealants
Brief Title: Effectiveness of Sealants on Molars
Acronym: sealants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 9500
Record Dates: First submitted 2016-09-06; First posted 2016-09-12 (Estimated); Last update posted 2022-08-11 (Actual); Status verified 2020-11

CONDITIONS: Tooth Decay
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: test and control tooth groups. Each patient is therefore his own witness
Who Masked: Participant
Masking Description: test and control tooth groups. Each patient is therefore his own witness
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- test tooth groups (Other): test tooth groups
  Interventions: Other: decayed tooth surfaces
- control tooth groups (Other): control tooth groups
  Interventions: Other: decayed tooth surfaces

INTERVENTIONS:
Other: decayed tooth surfaces — The main variable is the number of new decayed tooth surfaces between the end and the beginning of the research. The caries experience will also be evaluated and expressed by the index 'dmfs' (accumulation of decayed tooth surfaces over those missing or filled due to caries). The secondary variable will be the expression of the retention of AS. The comparison of caries incidence between the two groups of teeth (with and without AS) will take into account the membership of the teeth to the same subject by means of the statistical test Chi-McNemar two. Regression models logistics and Poisson regression will be used to test the effect of independent variables on the appearance of new cavities. The Stata statistical software will be used.

SUMMARY:
Currently, the real scope of sealants (AS) is poorly documented in temporary dentition and its effectiveness has not been demonstrated. Yet it seems reasonable that the AS in temporary dentition could slow the specific development of carious lesions in early childhood. In addition, this non-invasive approach could delay the conventional food and thus save financial costs for more complex treatments. Finally, the installation of AS could afford, as demonstrated in adult teeth, lowering the cariogenic bacteria prevalence engaged in the caries process.

DETAILED DESCRIPTION:
Currently, the real scope of sealants (AS) is poorly documented in temporary dentition and its effectiveness has not been demonstrated. Yet it seems reasonable that the AS in temporary dentition could slow the specific development of carious lesions in early childhood. In addition, this non-invasive approach could delay the conventional food and thus save financial costs for more complex treatments. Finally, the installation of AS could afford, as demonstrated in adult teeth, lowering the cariogenic bacteria prevalence engaged in the caries process.

Main objective: To evaluate the effect of AS on caries incidence in the deciduous dentition obtained over a period of three years, taking into account the risk of caries established initially.

Secondary objectives:

1. To assess the prevalence and caries attack sites at the end of each year
2. Estimate the retention rate (partial or complete) of the AS during the study
3. Determine the cost savings of treatment during the trial period

ELIGIBILITY:
Inclusion Criteria:

* Children who have at least two pairs (test / control) of healthy molars with occlusal surface or non cavitary initial injury.
* Children available for a follow-up 3 years
* Children being affiliated or beneficiary in a health insurance plan

Exclusion Criteria:

* Children involved in other research in the same field
* Child is exclusion period determined by previous research
* Children participating in research in the last three months its inclusion
* Parents do not understand French.
* Children deprived of liberty.
* Child participation Refusal
* Refusal to participate in either of the parents or legal representative

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
decayed tooth surfaces | 1 year
  The main variable is the number of new decayed tooth surfaces between the end and the beginning of the research. The caries experience will also be evaluated and expressed by the index 'dmfs' (accumulation of decayed tooth surfaces over those missing or filled due to caries). The secondary variable will be the expression of the retention of AS. The comparison of caries incidence between the two groups of teeth (with and without AS) will take into account the membership of the teeth to the same subject by means of the statistical test Chi-McNemar two. Regression models logistics and Poisson regression will be used to test the effect of independent variables on the appearance of new cavities. The Stata statistical software will be used.

SECONDARY OUTCOMES:
decayed tooth surfaces | 2 years
  The main variable is the number of new decayed tooth surfaces between the end and the beginning of the research. The caries experience will also be evaluated and expressed by the index 'dmfs' (accumulation of decayed tooth surfaces over those missing or filled due to caries). The secondary variable will be the expression of the retention of AS. The comparison of caries incidence between the two groups of teeth (with and without AS) will take into account the membership of the teeth to the same subject by means of the statistical test Chi-McNemar two. Regression models logistics and Poisson regression will be used to test the effect of independent variables on the appearance of new cavities. The Stata statistical software will be used.
decayed tooth surfaces | 3years
  The main variable is the number of new decayed tooth surfaces between the end and the beginning of the research. The caries experience will also be evaluated and expressed by the index 'dmfs' (accumulation of decayed tooth surfaces over those missing or filled due to caries). The secondary variable will be the expression of the retention of AS. The comparison of caries incidence between the two groups of teeth (with and without AS) will take into account the membership of the teeth to the same subject by means of the statistical test Chi-McNemar two. Regression models logistics and Poisson regression will be used to test the effect of independent variables on the appearance of new cavities. The Stata statistical software will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Estellle MOULIS, MCU-PH, Principal Investigator — University Hospital, Montpellier; olivier CHABADEL, MCU-PH, Principal Investigator — University Hospital, Montpellier
Locations (1):
- MOULIS, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chabadel O, Veronneau J, Montal S, Tramini P, Moulis E. Effectiveness of pit and fissure sealants on primary molars: A 2-yr split-mouth randomized clinical trial. Eur J Oral Sci. 2021 Feb;129(1):e12758. doi: 10.1111/eos.12758. Epub 2020 Dec 30. PMID 33377533